CLINICAL TRIAL: NCT02702024
Title: The Effectiveness of Double Incision Technique in Uterus Preserving Surgery for Placenta Percreta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Burak Yücel, Medical Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: DIforPP
Record Dates: First submitted 2016-02-26; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Placenta Percreta
Keywords: efficacy; double incision technique; uterus preserving surgery
MeSH Terms: conditions — Placenta Accreta

INTERVENTIONS:
Procedure: Double uterine incision technique in uterus preserving surgery for placenta percreta

SUMMARY:
Placenta percreta is a life-threatening condition that patients are under risk of massive bleeding. It readily necessitates very complicated surgery even leads to mortality. Cesarean hysterectomy is the procedure that is acknowledged worldwide, however, recent studies discussing conservative treatment with segmental resections were published. Fetal extraction and segmental resection could be performed from same (single uterine incision) or two different (double uterine incision) incisions. In this study, the investigators aimed to evaluate the effectiveness and the results of double uterine incision.

ELIGIBILITY:
Inclusion Criteria:

* Intraoperatively and pathologically confirmed diagnosis of placenta percreta

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Dates: Start 2014-01; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The success of segmental resection (Uterus preserving surgery) | Postoperative one month
  No need for hysterectomy due to massive hemorrhage or any other reason in postoperative one month

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Polat I, Yucel B, Gedikbasi A, Aslan H, Fendal A. The effectiveness of double incision technique in uterus preserving surgery for placenta percreta. BMC Pregnancy Childbirth. 2017 Apr 27;17(1):129. doi: 10.1186/s12884-017-1262-3. PMID 28449642